CLINICAL TRIAL: NCT02495857
Title: A Double-Blind, Randomized, Study of the Effectiveness and Safety of Hyaluronate Injectable Viscosupplement for Treatment of Osteoarthritis of the Knee
Brief Title: A Study of Hyaluronate Injectable Viscosupplement for Treatment of Osteoarthritis of the Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AV01.2015-0863
Record Dates: First submitted 2015-07-09; First posted 2015-07-13 (Estimated); Results first posted 2020-06-23 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Hyaluronate Injectable Viscosupplement (Experimental): Hyaluronate Injectable Viscosupplement (1% sodium hyaluronate). IA injection to the knee once weekly for 3 weeks
  Interventions: Device: Hyaluronate Injectable Viscosupplement
- Euflexxa IA injection (Active Comparator): Euflexxa IA injection to the knee once weekly for 3 weeks
  Interventions: Device: Euflexxa IA injection
- Placebo (Placebo Comparator): Placebo (normal saline). IA injection to the knee once weekly for 3 weeks
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Hyaluronate Injectable Viscosupplement — Test product of a 1% sodium hyaluronate for injection
  Other Names: 1% sodium hyaluronate
  Arms: Hyaluronate Injectable Viscosupplement
Device: Euflexxa IA injection — Brand product of a 1% sodium hyaluronate for injection
  Other Names: 1% sodium hyaluronate
  Arms: Euflexxa IA injection
Device: Placebo — 0.9% sodium chloride, sterile
  Other Names: Normal saline
  Arms: Placebo

SUMMARY:
The study is a prospective, multi-center, randomized, three-arm, parallel group, clinical study to evaluate the superiority of 3 weekly intra-articular (IA) doses of 2 mL of Investigational hyaluronate as compared to placebo injected into the target knee for the treatment of pain in subjects with Osteoarthritis (OA).The safety and effectiveness of the investigational product will also be compared with Euflexxa.

DETAILED DESCRIPTION:
The primary objective is to evaluate the safety and effectiveness of 3 weekly IA doses of 2 mL of hyaluronate viscosupplement as compared to placebo injected into the target knee for the treatment of pain in subjects with OA As secondary objectives, the study will evaluate the safety and effectiveness of 3 weekly IA doses of 2 mL of Viscosupplement as compared to Euflexxa injected into the target knee for the treatment of pain in subjects with OA. In addition, to assess the effect of Viscosupplement on pain, stiffness, and physical function of the target knee, as well as functional health and general well-being

ELIGIBILITY:
Inclusion Criteria:

* Chronic OA of target knee confirmed by American College of Rheumatology Criteria
* Pain due to OA in target knee that had been present for at least 6 months, with a moderate to severe pain score of >50 mm recorded on a 100 mm Visual Analogue Scale (VAS) following a 50-foot walk
* Subject agrees to discontinue all pain medications for at least 7 days prior to start of study
* A bilateral standing anteroposterior x-ray confirming Grade 2 or 3 OA of the target knee
* Body mass index ≤40kg/m2
* Able and willing to use only acetaminophen as the analgesic (rescue) study medication under the following conditions:

  * acetaminophen dose is not to exceed 4 grams (4000mg)/day
  * if the subject has known chronic liver disease, the maximum dose of acetaminophen is not to exceed 2 grams (2000 mg)/day
  * subject must be able and willing to discontinue acetaminophen at least 24 hours prior to all study-specific visits
* Ability to perform procedures required of the pain index evaluations (unassisted walking for a distance of 50 feet on a flat surface and going up and down stairs)
* Agrees to use a highly effective contraception
* Able and willing to complete effectiveness and safety questionnaires and able to read and understand study instructions

Exclusion Criteria:

* Any major injury to the target knee within the 12 months prior to the Screening and Enrollment Visit
* Any surgery to the target knee within the 12 months prior to the Screening and Enrollment Visit,
* Articular procedures such as transplants or ligament reconstruction to the target knee within 12 months prior to Screening and Enrollment Visit
* Inflammatory arthropathies such as rheumatoid arthritis, lupus arthropathy, or psoriatic arthritis
* Gout or calcium pyrophosphate diseases of the target knee that have flared within the 6 months prior to the Screening and Enrollment Visit
* X-ray findings of acute fractures, severe loss of bone density, avascular necrosis, and/or severe bone or joint deformity in the target knee
* Osteonecrosis of either knee
* Clinical signs and symptoms of active knee infection or crystal disease of the target knee
* Fibromyalgia, pes anserine bursitis, lumbar radiculopathy, and/or neurogenic or vascular claudication
* Significant anterior knee pain due to diagnosed isolated patella-femoral syndrome or chondromalacia in the target knee
* Significant target knee joint, infection or skin disorder infection within the 6 months prior to study enrollment
* Symptomatic OA of the hips, spine, or ankle, that interferes with the evaluation of the target knee
* Known hypersensitivity to acetaminophen or any of the study medications or their components
* Women of childbearing potential who are pregnant, nursing, or planning to become pregnant
* History of recurrent severe allergic or immune mediated reactions or other immune disorders
* Vascular insufficiency of lower limbs or peripheral neuropathy severe enough to interfere with the study evaluation
* Intra-arterial corticosteroid (investigational or marketed) in any joint within 3 months of Screening and Enrollment Visit
* Current treatment, or treatment within the 2 years prior to the Screening and Enrollment Visit, for any malignancy
* Active liver disease based on liver profile of aspartate aminotransferase, alanine aminotransferase, and conjugated bilirubin >2 times the upper limit of normal
* Renal insufficiency based on serum creatinine >2.0mg/dL
* Any intercurrent chronic disease or condition that might interfere with the completion of the study
* Current alcoholism and/or any known current addiction to pain medications
* Participation in any experimental device study within 6 months prior to the Screening and Enrollment Visit, or participation in an experimental drug study within 1 month prior to the Screening and Enrollment Visit.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 599 (Actual)
Dates: Start 2015-08-15 (Actual); Primary Completion 2016-12-05 (Actual); Study Completion 2016-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry Lay, PhD, Study Director — Actavis Inc.
Locations (2):
- United States (2):
  - Mehra, San Diego, California
  - Bretton, Albuquerque, New Mexico

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The populations for this study included the Safety Population, the modified Intent-to-Treat (mITT) population, and the Per-Protocol (PP) Population.
Groups:
- Hyaluronate Injectable Viscosupplement: Patients were administered intra-articular (IA) injection of 2 mL to the knee once weekly for 3 weeks.
- Euflexxa IA Injection: Patients received intra-articular (IA) injection of 2 mL to the knee once weekly for 3 weeks.
- Placebo Solution: Patients received intra-articular (IA) injection of 2mL to the knee once weekly for 3 weeks.
Period: Overall Study
Arm/Group | Hyaluronate Injectable Viscosupplement | Euflexxa IA Injection | Placebo Solution
Started | 200 | 200 | 199
Completed | 178 | 184 | 181
Not Completed | 22 | 16 | 18
Not completed — Adverse Event | 5 | 0 | 1
Not completed — Withdrawal by Subject | 9 | 6 | 10
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Protocol Violation | 1 | 1 | 2
Not completed — Lost to Follow-up | 4 | 5 | 3
Not completed — Other | 3 | 3 | 2

BASELINE CHARACTERISTICS:
Population: Intent to Treat Population
Groups:
- Generic Hyaluronate Injectable, 1%: Patients were administered intra-articular (IA) injection of 2 mL to the knee once weekly for 3 weeks.
- Euflexxa Injection 1%: Patients received intra-articular (IA) injection of 2 mL to the knee once weekly for 3 weeks.
- Vehicle Solution: Patients received intra-articular (IA) injection of 2mL to the knee once weekly for 3 weeks.
- Total: Total of all reporting groups
Arm/Group | Generic Hyaluronate Injectable, 1% | Euflexxa Injection 1% | Vehicle Solution | Total
Number analyzed (Participants) | 200 | 200 | 199 | 599
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (9.45) | 63.3 (9.36) | 62.0 (10.04) | 62.8 (9.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 83 | 89 | 251
  Male | 121 | 117 | 110 | 348
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 70 | 54 | 54 | 178
  Not Hispanic or Latino | 130 | 146 | 145 | 421
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 0 | 3
  Asian | 13 | 10 | 8 | 31
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 20 | 27 | 31 | 78
  White | 163 | 161 | 160 | 484
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the WOMAC Pain Score in the Target Knee at Week 26 [Western Ontario and McMaster Universities Arthritis Index (WOMAC®)]
Description: The primary effectiveness endpoint was the change from Baseline in the Western Ontario and McMaster Universities Arthritis Index (WOMAC®) pain score in the target knee at Week 26.The validated WOMAC was used to assess pain, stiffness, and physical function of the target knee.The range of pain score was 0 to 500 mm with higher scores for worse pain.
Time Frame: Baseline and 26 weeks
Population: Intention-To-Treat (ITT) Population
Measure: Mean (Standard Deviation); unit: Percentage of change from baseline
Arm/Group | Generic Hyaluronate Injectable, 1% | Euflexxa Injection 1% | Vehicle Solution
Number analyzed (Participants) | 200 | 200 | 199
Percentage of change from baseline | -51.43 (41.012) | -54.49 (37.042) | -36.86 (52.826)
Statistical Analysis 1: Comparison: Generic Hyaluronate Injectable, 1% vs Vehicle Solution; Test type: Superiority; Mean Difference (Net) = 36.18, 95% CI 2-sided [10.25 to 62.11]

2. Secondary Outcome: Change in Pain Over Time From Baseline to Week 1, Week 6, Week 12 and Week 26
Description: The change from Baseline in the WOMAC pain score over time (baseline to Week 1, Week 6, Week 12 and Week 26) using Western Ontario and McMaster Universities Arthritis Index (WOMAC®)].The validated WOMAC was used to assess pain, stiffness, and physical function of the target knee.The range of pain score was 0 to 500 mm with higher scores for worse pain.
Time Frame: 26 weeks
Population: Intention-To-Treat (ITT) Population
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | Generic Hyaluronate Injectable, 1% | Euflexxa Injection 1% | Vehicle Solution
Number analyzed (Participants) | 200 | 200 | 199
percentage of change from baseline
  Week 1 | -14.10 (30.568) | -15.13 (27.341) | -15.08 (32.680)
  Week 6 | -46.28 (41.042) | -49.91 (35.543) | -33.96 (68.782)
  Week 12 | -51.96 (40.894) | -52.47 (35.749) | -39.16 (58.080)
  Week 26 | -51.43 (41.012) | -54.49 (37.042) | -36.86 (52.826)
Statistical Analysis 1: Comparison: Generic Hyaluronate Injectable, 1% vs Euflexxa Injection 1%; Test type: Superiority; Mean Difference (Net) = 36.19, 95% CI 2-sided [10.25 to 62.11]

3. Secondary Outcome: Change in Stiffness of the Knee After 26 Weeks as Measured by the WOMAC Pain Score in the Target Knee at Week 26 [Western Ontario and McMaster Universities Arthritis Index (WOMAC®)]
Description: The change from baseline in the stiffness in the target knee at Week 26. The validated WOMAC was used to assess pain, stiffness, and physical function of the target knee.The range of stiffness score was 0 to 100 mm with higher scores for worse stiffness.
Time Frame: 26 weeks
Population: Intention-To-Treat (ITT) Population
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | Generic Hyaluronate Injectable, 1% | Euflexxa Injection 1% | Vehicle Solution
Number analyzed (Participants) | 200 | 200 | 199
percentage of change from baseline | -47.37 (45.275) | -47.25 (63.020) | -35.77 (63.103)
Statistical Analysis 1: Comparison: Generic Hyaluronate Injectable, 1% vs Euflexxa Injection 1%; Test type: Equivalence — From baseline to week 26 visit, change in the WOMAC stiffness score was evaluated; Mean Difference (Net) = 5.63, 95% CI 2-sided [-13.61 to 8.49]

ADVERSE EVENTS:
Time Frame: Data was collected for 26 weeks.
Groups:
- Euflexxa Injection 1%; Vehicle Solution: Patients were administered intra-articular (IA) injection of 2 mL to the knee once weekly for 3 weeks.
Arm/Group | Generic Hyaluronate Injectable, 1% | Euflexxa Injection 1% | Vehicle Solution
All-Cause Mortality (participants affected / at risk) | 0/199 | 0/199 | 0/197
Serious Adverse Events (participants affected / at risk) | 5/199 | 2/199 | 3/197
Other Adverse Events (participants affected / at risk) | 76/199 | 82/199 | 76/197
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Generic Hyaluronate Injectable, 1% (N=199) | Euflexxa Injection 1% (N=199) | Vehicle Solution (N=197)
Atrioventricular block complete (Cardiac disorders) | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Generic Hyaluronate Injectable, 1% (N=199) | Euflexxa Injection 1% (N=199) | Vehicle Solution (N=197)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 1
Meniere's disease (Ear and labyrinth disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 1 | 2 | 0
Conjunctivitis allergic (Eye disorders) | 1 | 0 | 0
Eyelid cyst (Eye disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Injection site joint pain (General disorders) | 5 | 1 | 12
Injection site joint effusion (General disorders) | 1 | 4 | 3
Injection site joint swelling (General disorders) | 1 | 2 | 3
Injection site pain (General disorders) | 2 | 2 | 1
Oedema peripheral (General disorders) | 2 | 1 | 2
Injection site erythema (General disorders) | 0 | 2 | 0
Injection site warmth (General disorders) | 0 | 2 | 0
Pain (General disorders) | 1 | 0 | 1
Asthenia (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 0
Injection site bruising (General disorders) | 0 | 0 | 1
Injection site haemorrhage (General disorders) | 0 | 0 | 1
Injection site reaction (General disorders) | 0 | 0 | 1
Injection site swelling (General disorders) | 0 | 0 | 1
Mass (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Swelling (General disorders) | 1 | 0 | 0
Tenderness (General disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 7 | 7 | 3
Nasopharyngitis (Infections and infestations) | 5 | 3 | 8
Bronchitis (Infections and infestations) | 5 | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 2 | 2
Sinusitis (Infections and infestations) | 0 | 3 | 1
Diverticulitis (Infections and infestations) | 1 | 1 | 0
Ear infection (Infections and infestations) | 0 | 2 | 0
Herpes zoster (Infections and infestations) | 2 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 1
Pharyngitis (Infections and infestations) | 1 | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 1 | 0
Bacterial infection (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 1 | 0
Epididymitis (Infections and infestations) | 0 | 1 | 0
Eye infection (Infections and infestations) | 0 | 0 | 1
Fungal infection (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Injection site infection (Infections and infestations) | 0 | 1 | 0
Oophoritis (Infections and infestations) | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 1 | 0
Parotitis (Infections and infestations) | 1 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 2 | 1 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Intervertebral disc injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Muscle injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood pressure increased (Investigations) | 1 | 1 | 0
Blood glucose increased (Investigations) | 0 | 1 | 0
Cardiac murmur (Investigations) | 0 | 1 | 0
Heart rate irregular (Investigations) | 0 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 | 26 | 24
Joint swelling (Musculoskeletal and connective tissue disorders) | 5 | 3 | 7
Joint crepitation (Musculoskeletal and connective tissue disorders) | 5 | 3 | 4
Joint effusion (Musculoskeletal and connective tissue disorders) | 4 | 2 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Plantar fascitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Joint instability (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Joint warmth (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Intraductal papilloma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Headache (Nervous system disorders) | 3 | 3 | 5
Presyncope (Nervous system disorders) | 1 | 0 | 2
Sciatica (Nervous system disorders) | 2 | 1 | 0
Sinus headache (Nervous system disorders) | 1 | 0 | 1
Balance disorder (Nervous system disorders) | 1 | 0 | 0
Cerebral small vessel ischaemic disease (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1
Renal pain (Renal and urinary disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the study may be published or presented by the Investigator(s) after the review by, and in consultation and agreement with the Sponsor, and such that confidential or proprietary information is not disclosed.